CLINICAL TRIAL: NCT01971320
Title: Evaluation of Transcutaneous Electrical Stimulation in Post Stroke Dysphagia
Acronym: TENSDEG
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/002/HP
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Oropharyngeal Dysphagia; Deglutition Disorders
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- active stimulation (Experimental): sensitive electrical stimulation applied during meals with Urostim I for 6 weeks
  Urostim I stimulation will be done during meals for 6 weeks
  Interventions: Device: Urostim I stimulation
- fake stimulation (Placebo Comparator): Urostim I stimulation will be done during meals for 6 weeks
  Fake sensitive electrical stimulation applied during meals with modified Urostim I who not deliver stimulation for 6 weeks
  Interventions: Device: Urostim I stimulation

INTERVENTIONS:
Device: Urostim I stimulation — Urostim I stimulation will be done during meals for 6 weeks

SUMMARY:
Oropharyngeal dysphagia induces aspirations which could be responsible of aspiration pneumonia and denutrition. It could be present in the majority of central neurological disease (degenerative or vascular disease), which explains that it is the first case of mortality in stroke. Two pilot studies realised by our research group aimed to demonstrate that sensitive transcutaneous electrical stimulation could improve swallowing coordination and reduce aspirations. This technique could be used at home.

The aim of this study is to demonstrate that sensitive electrical stimulation could improve oropharyngeal dysphagia in hemispheric stroke patients. 118 patients should be included in seven centers. Sensitive electrical stimulation will be applied either as active stimulation, either as a placebo. Active electrical stimulation will be realised at 80 hz during 30 minutes, under motor threshold and above sensitive threshold. It will be administrated via surface electrodes over the hyoid bone. Patients will be separated by randomisation.

Patients will be evaluated before and after 6 weeks of use. Methods will evaluation questionnaire, clinical examination and videofluoroscopy. The time of use will also be collected.

We wish to demonstrate that transcutaneous electrical stimulation is able to improve oropharyngeal dysphagia in stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* No contraindication to electrical stimulation
* Oropharyngeal dysphagia from 8 weeks diagnosed by videofluorosocpy with penetration aspiration scale > 3 or a residue ≥ 50%
* Due to an hemispheric stroke
* Patients able to understand the videofluroscopy and questionnaires
* For women in age of procreation, to have a contraception, a pregnacy test will be done if not
* Able to swallow (a nasogastric tube is not a contraindication to participate)

Exclusion Criteria:

* Pregnancy or breast feeding
* Psychiatric illnes
* Swallowing disorders before the stroke
* Contraindication to electrical stimulation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of oropharyngeal dysphagia symptoms | Week 6
  Evaluation of oropharyngeal dysphagia symptoms by questionnaire (dysphagia handicap index)

SECONDARY OUTCOMES:
Evaluation of oropharyngeal dysphagia symptoms | Week 6
  Evaluation of oropharyngeal dysphagia symptoms by videofluoroscopy and Swal-QoL questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eric VERIN, Professor, Principal Investigator — UH Rouen
Locations (6):
- France (6):
  - Centre les Herbiers, Bois-Guillaume
  - UH Bordeaux, Bordeaux
  - UH Limoges, Limoges
  - AP-HP Fernand WIDAL, Paris
  - UH Rouen, Rouen
  - UH Toulouse, Toulouse